CLINICAL TRIAL: NCT01065428
Title: Department of Critical Care Medicine, Nanjing Zhong-Da Hospital, Southeast University School of Medicine, China; Department of Critical Care Medicine St. Michaels's Hospital, University of Toronto, Canada
Brief Title: Extubation Readiness and Neuroventilatory Efficiency After Acute Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Ling Liu, Prof., Southeast University, China
Other Study IDs: 437129519
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Respiratory Failure
Keywords: neuromechanical efficiency; neuroventilatory efficiency; weaning; Respiration, Artificial
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Parameters of arterial blood gases, haemodynamic and mechanics of breathing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Weaning failure: Weaning failure:(1) failed SBT; (2) reintubation and /or resumption of support following successful extubation; or (3) die 48h following extubation.
- Weaning successful: Weaning successful:extubation and the absence of ventilatory support 48 h following the extubation

SUMMARY:
The aim of this study was to compare the indices of rapid shallow breathing, neuromechanical efficiency (NME), and neuroventilatory efficiency (NVE) between patients being successfully extubated and those who failed weaning.

DETAILED DESCRIPTION:
Patients, mechanically ventilated for > 24 h, were included when they met criteria for their first spontaneous breathing trial (SBT) on continuous positive airway pressure (CPAP) (5-6 cmH2O) for 30 minutes. Patients who did not fulfill the criteria for successful SBT, or required assist, or deceased within 48h post-extubation were considered extubation failure (F). Patients who completed the SBT and remained extubated > 48 h were considered successfully extubated (S). Before and during the SBT, arterial blood gases, heart, rate, blood pressure, and EAdi, flow, Vt, f, and, airway pressure (Paw) were measured. At 0, 5, 10, 15 and 30 minutes of the SBT, f/Vt, diaphragm electrical activity (EAdi), NME, and NVE were calculated. NME was calculated as Paw/EAdi during inspiratory occlusion. NVE was calculated as Vt/EAdi during unassisted inspirations.Arterial blood gases, heart rate, and blood pressure were measured. The receiver operating characteristic (ROC) curve was calculated to evaluate the predictive performance of each index.

ELIGIBILITY:
Inclusion Criteria:

* We chose a number of eligible patients which were admitted to ICU of the Zhong-Da Hospital and required mechanical ventilation for more than 24 h.

Exclusion Criteria:

(1) age <18 or >85 years, (2) tracheostomy, (3) treatment abandonment, (4) history of esophageal varices, (5) gastro-esophageal surgery in the previous 12 months or gastro-esophageal bleeding in the previous 30 days, (6) coagulation disorders (INR ratio>1.5 and APTT>44 s), (7) history of acute central or peripheral nervous system disorder or severe neuromuscular disease, (8) history of leukemia, severe chronic liver or chronic cardiac disease, (9) solid organ transplantation, (10) malignant tumor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who required mechanical ventilation for more than 24 h.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, MD, Phd, Study Director — Southeast University
Locations (1):
- Nanjing Zhong-Da Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Liu L, Liu H, Yang Y, Huang Y, Liu S, Beck J, Slutsky AS, Sinderby C, Qiu H. Neuroventilatory efficiency and extubation readiness in critically ill patients. Crit Care. 2012 Jul 31;16(4):R143. doi: 10.1186/cc11451. PMID 22849707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In a 20 beds general ICU of a teaching hospital, from December 2008 to May 2010, 52 patients , mechanically ventilated for > 24 h, were included when they deemed ready for extubation by the clinical team and fulfilled established weaning criteria.
Pre-assignment Details: Nasogastric tube Eligible patient was replaced with a modified EAdi catheter (Maquet, Solna, Sweden). Then the patients were switched to a Servo-i ventilator capable of processing signals of EAdi automatically.
Groups:
- Weaning Failure: Weaning failure:(1) failed spontaneous breathing trials (SBT); (2) reintubation and /or resumption of support following successful extubation; or (3) die 48h following extubation.
Period: Overall Study
Arm/Group | Weaning Failure | Weaning Successful
Started | 17 | 35
Completed | 17 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weaning Failure | Weaning Successful | Total
Number analyzed (Participants) | 17 | 35 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 13 | 14
  >=65 years | 16 | 22 | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 76.0 (6.4) | 65.2 (18.5) | 68.8 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 8 | 24 | 32
Region of Enrollment [Number; unit: participants]
  China | 17 | 35 | 52

OUTCOME MEASURES:

1. Primary Outcome: Neuroventilatory Efficiency (NVE)
Description: NVE is the ratio of tidal volume and diaphragm electrical activity (Vt/EAdi).It is a value describing how effective a patient's breathing is.
Time Frame: at 30 minutes of the spontaneous breathing trials (SBT)
Measure: Mean (Standard Deviation); unit: ml/uV
Arm/Group | Weaning Failure | Weaning Successful
Number analyzed (Participants) | 17 | 35
ml/uV | 17.6 (10.7) | 39.9 (23.9)
Statistical Analysis 1: Comparison: Weaning Failure vs Weaning Successful; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Neuromechanical Efficiency (NME)
Description: NME is the ratio between inspiratory pressure generation and EAdi (Paw/EAdi).
Time Frame: at 30 minutes of the spontaneous breathing trials (SBT)
Measure: Mean (Standard Deviation); unit: cmH2O/uV
Arm/Group | Weaning Failure | Weaning Successful
Number analyzed (Participants) | 17 | 35
cmH2O/uV | 1.13 (0.71) | 1.77 (0.79)
Statistical Analysis 1: Comparison: Weaning Failure vs Weaning Successful; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During the 30 nints of SBT, and 48 hours after extubation
Description: There was no additional intervention being used in this observational study. We just observed the NVE and NME during a local protocol of SBT and weaning. In addition to the risk caused by the routine SBT and weaning, there was no additional risk during the observation period.
Arm/Group | Weaning Failure | Weaning Successful
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/35
Other Adverse Events (participants affected / at risk) | 0/17 | 0/35

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No